CLINICAL TRIAL: NCT03873545
Title: A Prospective, Multi-Center Study Evaluating ProChondrix® CR for the Repair of Focal Articular Cartilage Defects in the Knee
Brief Title: Prospective Evaluation of ProChondrix CR for Repair of Articular Cartilage Defects on Femoral Condyle and Patella
Status: Active, not recruiting | Type: Observational
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-002
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cartilage Injury; Cartilage Damage
Keywords: Cartilage; Cartilage Injury; Cartilage Repair; Cartilage Damage; Cartilage Lesion; Cartilage Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cryopreserved Osteochondral Allograft — This tissue is a laser-etched, cryopreserved fresh osteochondral allograft that was developed as a single-stage alternative for articular cartilage restoration.
  Other Names: ProChondrix CR

SUMMARY:
The purpose of this clinical study is to evaluate the use of ProChondrix Cryopreserved Osteochondral Allograft to obtain evidence of effectiveness, defined as an improvement in physical function and pain, when used on a symptomatic cartilage defect on the femoral condyle or patella in a mechanically stable knee.

DETAILED DESCRIPTION:
This clinical study will use a multi-center, prospective design, to evaluate ProChondrix CR in approximately 80 patients who are scheduled to undergo treatment of a cartilage defect on the femoral condyle or patella.Patient follow-up will include a period of 60 months after surgery. During this follow-up period, each patient will be evaluated seven (7) times at: 3, 6, 12, 24, 36, 48 and 60 months after surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 and ≤ 60 years old at the time of surgery;
* Symptomatic patient presenting with moderate to severe pain in the index knee - unresponsive to conservative treatment (i.e. medication, bracing, physical therapy) and/or previous surgical intervention;
* Radiographically diagnosed, by MRI, or through arthroscopy, to have a cartilage defect on the femoral condyle or patella between ≥ 1 cm2 and ≤ 5 cm2, measured as a rectangle length x width;
* Will be having a marrow stimulation plus ProChondrix CR procedure;
* Has an intact meniscus (maximum of ≤50% resected);
* Have the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.

Exclusion Criteria:

* Has > 5° of varus or valgus deformity;
* Bipolar articular cartilage involvement (kissing lesions) of the ipsilateral compartment (i.e. > than ICRS Grade 2 on the opposing articular surface);
* Associated damage to the underlying subchondral bone >2 mm requiring osseous repair;
* Requires concomitant ligament repair other than Anterior Cruciate Ligament (ACL) or Medial Patella-Femoral Ligament (MPFL) reconstruction;
* Body Mass Index (BMI)of ≥ 35 kg/m2;
* Active malignancy: undergoing treatment for tumor or boney traumatic injury or a history of any invasive malignancy (except non-melanoma skin cancer), unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
* Clinical and/or radiographic disease in the affected joint that includes: osteoarthritis or avascular necrosis, gout or a history of gout or pseudogout, osteochondritis dissecans with significant bone loss;
* Cartilage lesion location such that the implanted graft will not be adequately shouldered;
* Active local microbial infection or a systemic infection, including prior or pending treatment for HIV, syphilis, Hepatitis B or Hepatitis C;
* Currently immunologically suppressed or immunocompromised, or a medical condition requiring radiation, chemotherapy or immunosuppression;
* Unstable cardiovascular, renal, hepatic, endocrine and/or pulmonary disease, cancer or uncontrolled diabetes;
* Has a history of any inflammatory or connective tissue disease, such as, systemic lupus erythematosus (SLE), Addison's disease, Crohn's disease, multiple sclerosis, polychondritis or rheumatoid arthritis;
* Received hyaluronic acid injections into the joint space ≤ 90 days prior to surgery;
* Is a female patient who is pregnant;
* Physically or mentally compromised (i.e. being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease) in a manner that would compromise his/her ability to participate in the clinical study;
* Has a history of substance abuse (recreational drugs, alcohol) or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an in-patient substance abuse program;
* Patients who, in the opinion of the Investigator, would not be able or willing to comply with the protocol;
* Is currently involved in a study of another investigational product for similar purpose or has been in the previous 90 days;
* Has any contraindications for MRI;
* Is a ward of the state, prisoner, or transient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Skeletally mature patients between the ages of ≥18 and ≤ 60 who have a symptomatic cartilage defect (Grade 3 or 4) on the femoral condyle or patella, in a mechanically stable knee, or is being mechanically stabilized in the same procedure, between ≥ 1 cm2 and ≤ 5 cm2, measured as a rectangle length x width, as confirmed by MRI or arthroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective International Knee Documentation Committee (IKDC) Score | Baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Change in physical pain and function as assessed by IKDC score from baseline to 60 months post-surgery

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Change of physical pain as assessed by KOOS score from baseline to 60 months post-surgery
SF-12 survey | Baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Change in functional health and well-being as assessed by SF-12 survey from baseline to 60 months post-surgery
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Scores | 12, 24 and 60 months
  Assessment of repair cartilage structure

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Beacon Orthopaedics & Sports Medicine, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No